CLINICAL TRIAL: NCT00635817
Title: A Phase 3, Randomized, Multi-Center, Open-Label Study to Evaluate the Efficacy and Safety of Leuprolide Acetate 11.25 and 30 mg Formulations in Children With Central Precocious Puberty
Brief Title: A Study of Leuprolide 11.25 mg and 30 mg Administered Every 3 Months to Treat Central Precocious Puberty
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: L-CP07-167
Record Dates: First submitted 2008-03-07; First posted 2008-03-14 (Estimated); Results first posted 2011-02-09 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-10

CONDITIONS: Puberty, Precocious
Keywords: CPP; central precocious puberty; pediatrics; suppression of luteinizing hormone; Lupron; leuprolide acetate; depot formulation; GnRHa; GnRH agonist; GnRH analog; luteinizing hormone
MeSH Terms: conditions — Puberty, Precocious | interventions — Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Leuprolide acetate 11.25 mg (Experimental): There are 2 arms that received leuprolide acetate 11.25 mg. Subjects who are treatment naive to leuprolide acetate are designated to be in Arm A and subjects who have previously been treated with leuprolide acetate are designated to be in Arm B.
  Interventions: Drug: Leuprolide acetate 11.25 mg
- Leuprolide acetate 30 mg (Experimental): There are 2 arms that received leuprolide acetate 30 mg. Subjects who are treatment naive to leuprolide acetate are designated to be in Arm C and subjects who have previously been treated with leuprolide acetate are designated to be in Arm D.
  Interventions: Drug: Leuprolide acetate 30 mg

INTERVENTIONS:
Drug: Leuprolide acetate 11.25 mg — Two intramuscular injections of leuprolide acetate for depot suspension 11.25 mg administered 3 mo apart.
  Other Names: ABT-818; leuprolide acetate; Lupron
  Arms: Leuprolide acetate 11.25 mg
Drug: Leuprolide acetate 30 mg — Two intramuscular injections of leuprolide acetate for depot suspension 30 mg administered 3 mo apart.
  Other Names: ABT-818; leuprolide acetate; Lupron
  Arms: Leuprolide acetate 30 mg

SUMMARY:
The purpose of this study is to determine if 11.25 and 30 mg formulations of leuprolide are effective in treating children with Central Precocious Puberty (CPP).

DETAILED DESCRIPTION:
Study Design:

A total of 80 children with confirmed CPP were planned to be enrolled and randomized in a 1:1 ratio to receive 2 injections of either leuprolide acetate 11.25 mg or 30 mg depot formulation, each injection administered 3 mo apart (6 mo of treatment):

This study includes a 4-week Screening Period, two 3-mo treatment cycles, and a posttreatment follow-up period (12 weeks following the Mo 6 visit). Study visits will occur at Screening, Day 1, Week 2 (only for subjects participating in the pharmacokinetic subset), Mo 1, 2, 3, Mo 6/Early Termination, and 12 weeks later, for the Posttreatment Follow-up Visit.

This study was conducted at 18 sites in the United States and 4 sites in Puerto Rico.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a clinical diagnosis of CPP.
* Eligible to receive at least 6 mo of therapy to treat CPP after study entry.
* Bone age advanced at least 1 year beyond the chronological age at time of diagnosis or first treatment.
* In general good health with no uncontrolled, clinically significant disease which would interfere with bone maturation or mask the objectives of this protocol as assessed by the investigator.

Additional criteria for subjects who have not had previous treatment:

* Girls 2-8 years inclusive or Boys 2-9 years inclusive at Day 1.
* Has pretreatment pubertal response to leuprolide acetate stimulation (luteinizing hormone ≥8 mIU/mL) at Screening.
* Breast pubertal staging of at least 2 in girls; testicular volume of at least 4 cc or testicular length greater than 2.5 cm in boys at Screening.

Additional criteria for subjects previously treated:

* Girls 2-10 years inclusive or boys 2-11 years inclusive at Day 1.
* Must have been on standard gonadotropin releasing hormone analog therapy for at least the 6 mo prior to Day 1.
* Has documented maintenance of luteinizing hormone suppression as evidenced by peak stimulated level <4 mIU/mL at Screening.

Exclusion Criteria:

* Incomplete precocious puberty (premature thelarche, premature adrenarche).
* Peripheral precocious puberty: gonadal or adrenal tumors, congenital adrenal hyperplasia, testotoxicosis in boys, human chorionic gonadotropin secreting tumor or McCune-Albright syndrome in girls.
* Evidence of any abnormal pituitary, hypothalamic, adrenal, thyroid and gonadal function other than premature secretion of gonadotropins not adequately controlled.
* Unstable intracranial tumors (unresponsive to treatment/expanding) except hamartoma.
* Previous treatment with GnRHa therapy requiring leuprolide acetate for depot suspension >15 mg monthly.
* Bone age >13 years for girls and >14 years for boys.
* Any other condition interfering with growth, ie, skeletal dysplasia, cerebral palsy.
* Chronic illness requiring treatment that may interfere with growth, ie, chronic steroid use, renal failure, moderate to severe scoliosis.
* Diagnosis of short stature, ie more than 2.25 standard deviations below the mean height for age (growth chart measurement).
* Prior or current therapy with medroxyprogesterone acetate or growth hormone.
* Has an abnormal laboratory value suggesting a clinically significant underlying disease .
* Creatinine >1.5 mg/dL, alanine aminotransferase and/or aspartate aminotransferase >2.0 x upper limit of normal, or total bilirubin >2.0 mg/dL with aspartate aminotransferase/alanine aminotransferase elevated above normal limits.
* Positive pregnancy test.
* Known hypersensitivity to study medication or its excipients.
* Participation in another drug research within 3 mo of enrollment into this study.
* Prior or current therapy with insulin-like growth factor-1.
* Use of an estrogen preparation within 2 mo prior to Day 1.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2008-06; Primary Completion 2010-01 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bacher, MD,, Study Director — Abbott
Locations (25):
- United States (21):
  - Site Reference ID/Investigator# 8765, Birmingham, Alabama
  - Site Reference ID/Investigator# 11522, Long Beach, California
  - Site Reference ID/Investigator# 8756, Los Angeles, California
  - Site Reference ID/Investigator# 8755, San Diego, California
  - Site Reference ID/Investigator# 8761, San Diego, California
  - Site Reference ID/Investigator# 8772, Stanford, California
  - Site Reference ID/Investigator# 8749, Greenwood Village, Colorado
  - Site Reference ID/Investigator# 8771, Gainesville, Florida
  - Site Reference ID/Investigator# 8764, Jacksonville, Florida
  - Site Reference ID/Investigator# 17621, Pensacola, Florida
  - Site Reference ID/Investigator# 8752, Indianapolis, Indiana
  - Site Reference ID/Investigator# 8766, Shreveport, Louisiana
  - Site Reference ID/Investigator# 8768, Minneapolis, Minnesota
  - Site Reference ID/Investigator# 17341, Saint Paul, Minnesota
  - Site Reference ID/Investigator# 8759, Kansas City, Missouri
  - Site Reference ID/Investigator# 8750, Oklahoma City, Oklahoma
  - Site Reference ID/Investigator# 8760, Tulsa, Oklahoma
  - Site Reference ID/Investigator# 8763, Hershey, Pennsylvania
  - Site Reference ID/Investigator# 8754, Salt Lake City, Utah
  - Site Reference ID/Investigator# 8762, Seattle, Washington
  - Site Reference ID/Investigator# 8753, Seattle, Washington
- Puerto Rico (4):
  - Site Reference ID/Investigator# 17922, Bayamón
  - Site Reference ID/Investigator# 17923, Ponce
  - Site Reference ID/Investigator# 18242, San Juan
  - Site Reference ID/Investigator# 19661, San Juan

REFERENCES:
- [Derived] Lee PA, Klein K, Mauras N, Neely EK, Bloch CA, Larsen L, Mattia-Goldberg C, Chwalisz K. Efficacy and safety of leuprolide acetate 3-month depot 11.25 milligrams or 30 milligrams for the treatment of central precocious puberty. J Clin Endocrinol Metab. 2012 May;97(5):1572-80. doi: 10.1210/jc.2011-2704. Epub 2012 Feb 16. PMID 22344198

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eighteen sites in the US and 4 sites in Puerto Rico enrolled subjects into the study. The first subject was randomized 17 June 2008 and the last subject was randomized 12 Aug 2009.
Pre-assignment Details: Subjects were randomized in a 1:1 ratio to 1 of the 2 treatment arms. To ensure balanced randomization, the study drug assignment was stratified on the basis of whether subjects were treatment-naive or had been treated with GnRHa previously.
Groups:
- Leuprolide Acetate 11.25 mg - Treatment Naive; Leuprolide Acetate 11.25 mg - Previous Treatment; Leuprolide Acetate 30 mg - Treatment Naive; Leuprolide Acetate 30 mg - Previous Treatment: Subjects who received at least 1 dose of study drug.
Period: Overall Study
Arm/Group | Leuprolide Acetate 11.25 mg - Treatment Naive | Leuprolide Acetate 11.25 mg - Previous Treatment | Leuprolide Acetate 30 mg - Treatment Naive | Leuprolide Acetate 30 mg - Previous Treatment
Started | 21 | 21 | 21 | 21
Completed | 15 | 19 | 19 | 21
Not Completed | 6 | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Leuprolide Acetate 11.25 mg - Treatment Naive | Leuprolide Acetate 11.25 mg - Previous Treatment | Leuprolide Acetate 30 mg - Treatment Naive | Leuprolide Acetate 30 mg - Previous Treatment | Total
Number analyzed (Participants) | 21 | 21 | 21 | 21 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 21 | 21 | 21 | 21 | 84
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: Years] | 7.4 (1.47) | 8.1 (1.83) | 7.3 (1.74) | 8.4 (1.75) | 7.8 (1.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 20 | 19 | 18 | 76
  Male | 2 | 1 | 2 | 3 | 8
Region of Enrollment [Number; unit: Participants]
  North America | 21 | 21 | 21 | 21 | 84

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Suppression of Peak Stimulated Luteinizing Hormone (<4 mIU/mL) From Month 2 Through Month 6
Description: Percentage of participants with suppression of peak stimulated luteinizing hormone that was measured after a gonadotropin-releasing hormone agonist (GnRHa) stimulation test at Month (Mo) 2, 3, and 6. The analysis was performed according to a life table method. Subjects who withdrew without peak-stimulated luteinizing hormone >= 4 mIU/mL were censored at their last measurement of peak-stimulated luteinizing hormone.
Time Frame: Month 2 through 6
Population: Subjects must have received at least 1 dose of study drug and had at least 1 postbaseline measurement of peak stimulated luteinizing hormone at Mo 2 or afterward defined as the intent-to-treat population.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Leuprolide Acetate 11.25 mg - Treatment Naive | Leuprolide Acetate 11.25 mg - Previous Treatment | Leuprolide Acetate 30 mg - Treatment Naive | Leuprolide Acetate 30 mg - Previous Treatment
Number analyzed (Participants) | 21 | 21 | 21 | 21
Percentage of Participants | 76.2 (9.29) [58.0 to 94.4] | 80.7 (8.69) [63.6 to 97.7] | 90.5 (6.41) [77.9 to 100] | 100 (0.00) [100 to 100]

2. Secondary Outcome: Percentage of Participants With Suppression of Basal Estradiol <20 pg/mL by Visit
Description: Percentage of participants with suppression of estradiol, out of the number of girls with at least 1 estradiol measurement at each visit (n/N%). Only girls are analyzed in this outcome measure. Observed data were used with no imputation for missing data.
Time Frame: Month 1, 2, 3 and 6
Population: Subjects must have received at least 1 dose of study drug and had at least 1 postbaseline measurement defined as the intent-to-treat population.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Leuprolide Acetate 11.25 mg - Treatment Naive | Leuprolide Acetate 11.25 mg - Previous Treatment | Leuprolide Acetate 30 mg - Treatment Naive | Leuprolide Acetate 30 mg - Previous Treatment
Number analyzed (Participants) | 19 | 20 | 19 | 18
Percentage of Participants
  Mo 1 (Arm A N=17, B N=18, C N=19, D N=16) | 100 [80.5 to 100] | 100 [81.5 to 100] | 100 [82.4 to 100] | 100 [79.4 to 100]
  Mo 2 (Arm A N=19, B N=14, C N=19, D N=14) | 94.7 [74.0 to 99.9] | 100 [76.8 to 100] | 100 [82.4 to 100] | 100 [76.8 to 100]
  Mo 3 (Arm A N=15, B N=18, C N=17, D N=18) | 100 [78.2 to 100] | 100 [81.5 to 100] | 100 [80.5 to 100] | 100 [81.5 to 100]
  Mo 6 (Arm A N=12, B N=16, C N=15, D N=17) | 100 [73.5 to 100] | 93.8 [69.8 to 99.8] | 100 [78.2 to 100] | 100 [80.5 to 100]

3. Secondary Outcome: Percentage of Participants With Suppression of Testosterone in <30 ng/dL by Visit
Description: Percentage of participants with suppression of testosterone, out of the number of boys with at least 1 testosterone measurement at each visit (n/N%). Only boys are analyzed in this outcome measure. Observed data were used with no imputation for missing data.
Time Frame: Month 1, 2, 3 and 6
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Leuprolide Acetate 11.25 mg - Treatment Naive | Leuprolide Acetate 11.25 mg - Previous Treatment | Leuprolide Acetate 30 mg - Treatment Naive | Leuprolide Acetate 30 mg - Previous Treatment
Number analyzed (Participants) | 2 | 1 | 2 | 3
Percentage of Participants
  Mo 1 (Arm A N=2, B N=1, C N=2, D N=3) | 50.0 [1.3 to 98.7] | 100 [2.5 to 100] | 100 [15.8 to 100] | 100 [29.2 to 100]
  Mo 2 (Arm A N=2, B N=1, C N=2, D N=3) | 50.0 [1.3 to 98.7] | 100 [2.5 to 100] | 100 [15.8 to 100] | 100 [29.2 to 100]
  Mo 3 (Arm A N=2, B N=1, C N=2, D N=3) | 50.0 [1.3 to 98.7] | 100 [2.5 to 100] | 100 [15.8 to 100] | 100 [29.2 to 100]
  Mo 6 (Arm A N=1, B N=1, C N=2, D N=3) | 100 [2.5 to 100] | 100 [2.5 to 100] | 100 [15.8 to 100] | 100 [29.2 to 100]

4. Secondary Outcome: Peak-stimulated Luteinizing Hormone Concentration by Visit
Description: Observed data were used with no imputation for missing data.
Time Frame: Baseline, Month 1, 2, 3 and 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | Leuprolide Acetate 11.25 mg - Treatment Naive | Leuprolide Acetate 11.25 mg - Previous Treatment | Leuprolide Acetate 30 mg - Treatment Naive | Leuprolide Acetate 30 mg - Previous Treatment
Number analyzed (Participants) | 21 | 21 | 21 | 21
mIU/mL
  Baseline (Arm A N=21, B N=21, C N=21, D N=21) | 45.9 (42.38) | 1.8 (1.78) | 23.5 (16.76) | 1.7 (1.09)
  Mo 1 (Arm A N=21, B N=21, C N=21, D N=21) | 4.4 (7.29) | 1.7 (1.36) | 1.9 (1.74) | 1.4 (0.76)
  Mo 2 (Arm A N=21, B N=20, C N=21, D N=20) | 4.5 (7.20) | 2.0 (1.48) | 2.0 (2.25) | 1.5 (0.73)
  Mo 3 (Arm A N=16, B N=20, C N=20, D N=21) | 2.3 (1.23) | 1.8 (1.10) | 1.4 (0.78) | 1.5 (0.61)
  Mo 6 (Arm A N=15, B N=18, C N=18, D N=21) | 2.0 (0.85) | 2.5 (2.43) | 1.6 (0.95) | 1.5 (0.89)

5. Secondary Outcome: Percentage of Participants With Suppression of the Physical Signs of Puberty (Breast Development) at Month 6
Description: Percentage of participants with suppression of breast development, out of the number of girls with pubertal staging of breast development (n/N%). Only girls are analyzed in this outcome measure. Breast development was rated from Stage 1 (early development) through Stage 5 (full development) according to a Tanner Staging pictogram. Girls entering the study with fully developed breasts (Stage 5) were excluded from this analysis. Observed data were used with no imputation for missing data.
Time Frame: Month 6
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Leuprolide Acetate 11.25 mg - Treatment Naive | Leuprolide Acetate 11.25 mg - Previous Treatment | Leuprolide Acetate 30 mg - Treatment Naive | Leuprolide Acetate 30 mg - Previous Treatment
Number analyzed (Participants) | 14 | 18 | 17 | 17
Percentage of Participants | 92.9 [66.1 to 99.8] | 88.9 [65.3 to 98.6] | 82.4 [56.6 to 96.2] | 82.4 [56.6 to 96.2]

6. Secondary Outcome: Percentage of Participants With Suppression of the Physical Signs of Puberty (Testicular Volume and Genital Development) at Month 6
Description: Percentage of participants with suppression of genital development and testicular volume, out of the number of boys with pubertal staging of genital development or testicular volume (n/N%). Only boys are analyzed in this outcome measure. External genital development (testes and penis) was rated from Stage 1 (early development) through Stage 5 (full development) according to a Tanner Staging pictogram. Boys entering the study with fully developed genitals (Stage 5) were excluded from this analysis. Observed data were used with no imputation for missing data.
Time Frame: Month 6
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Leuprolide Acetate 11.25 mg - Treatment Naive | Leuprolide Acetate 11.25 mg - Previous Treatment | Leuprolide Acetate 30 mg - Treatment Naive | Leuprolide Acetate 30 mg - Previous Treatment
Number analyzed (Participants) | 1 | 1 | 2 | 3
Percentage of Participants | 100 [2.5 to 100] | 0 [0.0 to 97.5] | 50 [1.3 to 98.7] | 33.3 [0.8 to 90.6]

7. Secondary Outcome: Change From Baseline in Incremental Growth Rate (cm/Year) at Month 6
Description: The growth rate at baseline was the growth rate during the last year before the start of treatment and was calculated with the measurement closest to Day -336 (before Day -30) and the measurement up to Day 1. Growth rate at Month 6 was defined as the ratio of the change in height from Day 1 to the change in chronological age, with an approximate 6-month interval between the 2 height measurements. Observed data were used with no imputation for missing data.
Time Frame: Baseline and Month 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | Leuprolide Acetate 11.25 mg - Treatment Naive | Leuprolide Acetate 11.25 mg - Previous Treatment | Leuprolide Acetate 30 mg - Treatment Naive | Leuprolide Acetate 30 mg - Previous Treatment
Number analyzed (Participants) | 20 | 21 | 21 | 21
cm/year
  Baseline (Arm A N=20, B N=21, C N=21, D N=21) | 7.25 (5.30) | 6.58 (2.39) | 7.83 (5.96) | 6.05 (1.55)
  Mo 6 (Arm A N=14, B N=19, C N=19, D N=21) | -2.51 (5.29) | -0.98 (2.24) | -2.34 (4.22) | -0.91 (2.45)
Statistical Analysis 1: Comparison: Leuprolide Acetate 11.25 mg - Treatment Naive; Summary statistics were calculated and tests of significance of the change versus no change were performed; Test type: Superiority or Other; p = 0.099, t-test, 2 sided — There were no adjustments for multiple comparisons
Statistical Analysis 2: Comparison: Leuprolide Acetate 11.25 mg - Previous Treatment; Summary statistics were calculated and tests of significance of the change versus no change were performed; Test type: Superiority or Other; p = 0.074, t-test, 2 sided — There were no adjustments for multiple comparisons
Statistical Analysis 3: Comparison: Leuprolide Acetate 30 mg - Treatment Naive; Summary statistics were calculated and tests of significance of the change versus no change were performed; Test type: Superiority or Other; p = 0.026, t-test, 2 sided — There were no adjustments for multiple comparisons
Statistical Analysis 4: Comparison: Leuprolide Acetate 30 mg - Previous Treatment; Summary statistics were calculated and tests of significance of the change versus no change were performed; Test type: Superiority or Other; p = 0.102, t-test, 2 sided — There were no adjustments for multiple comparisons

8. Secondary Outcome: Ratio of Change From Baseline in Bone Age/Change From Baseline in Chronological Age at Month 6
Description: The ratio at Month 6 was calculated as (bone age at Month 6 - bone age at baseline)/(chronological age at Month 6 - chronological age at baseline). Observed data were used with no imputation for missing data. Baseline bone-age radiograph was performed at or within 3 months of the Screening Visit.
Time Frame: Baseline to Month 6
Population: Participants must have received at least 1 dose of study drug and had at least 1 postbaseline measurement defined as the intent-to-treat population.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Leuprolide Acetate 11.25 mg - Treatment Naive | Leuprolide Acetate 11.25 mg - Previous Treatment | Leuprolide Acetate 30 mg - Treatment Naive | Leuprolide Acetate 30 mg - Previous Treatment
Number analyzed (Participants) | 15 | 18 | 18 | 21
Ratio | 0.59 (0.59) | 0.50 (0.57) | 1.00 (0.74) | 1.07 (1.60)
Statistical Analysis 1: Comparison: Leuprolide Acetate 11.25 mg - Treatment Naive; Summary statistics were calculated and tests of significance of the ratio versus 1 were performed. All analyses and summaries were conducted separately for the 2 treatment groups (subjects who received leuprolide acetate depot 11.25 mg and 30 mg); Test type: Superiority or Other; p = 0.008, Wilcoxon (Mann-Whitney) — There were no adjustments for multiple comparisons
Statistical Analysis 2: Comparison: Leuprolide Acetate 11.25 mg - Previous Treatment; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.002, Wilcoxon (Mann-Whitney) — There were no adjustments for multiple comparisons
Statistical Analysis 3: Comparison: Leuprolide Acetate 30 mg - Treatment Naive; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.347, Wilcoxon (Mann-Whitney) — There were no adjustments for multiple comparisons
Statistical Analysis 4: Comparison: Leuprolide Acetate 30 mg - Previous Treatment; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.150, Wilcoxon (Mann-Whitney) — There were no adjustments for multiple comparisons

9. Post Hoc Outcome: Percentage of Participants With Suppression of Peak Stimulated Luteinizing Hormone (< 4 mIU/mL) From Month 2 Through Month 6 (Simple Percentage With Binomial Exact Confidence Intervals)
Description: Percentage of participants with suppression of peak stimulated luteinizing hormone that was measured after a GnRHa stimulation test at Mo 2, 3, and 6. A simple percentage and binomial exact confidence intervals were used in this analysis. Participants who withdrew with luteinizing hormone that remained suppressed were counted as a success. This analysis was performed after the clinical study report was completed and is included to match the FDA package insert.
Time Frame: Month 2 through 6
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Leuprolide Acetate 11.25 mg - Treatment Naive | Leuprolide Acetate 11.25 mg - Previous Treatment | Leuprolide Acetate 30 mg - Treatment Naive | Leuprolide Acetate 30 mg - Previous Treatment
Number analyzed (Participants) | 21 | 21 | 21 | 21
Percentage of Participants | 76.2 [52.8 to 91.8] | 81.0 [58.1 to 94.6] | 90.5 [69.6 to 98.8] | 100.0 [83.9 to 100.0]

10. Post Hoc Outcome: Percentage of Participants With a Decrease From Baseline in the Ratio of Bone Age to Chronological Age at Month 6 Compared to Baseline
Description: The ratio at baseline or Month 6 was calculated as bone age at baseline or Month 6/chronological age at baseline or Month 6. The percentage of participants with a decrease in the ratio was calculated as a simple percentage for each dose group. Observed data were used with no imputation for missing data. The baseline time frame was increased from the secondary outcome in this analysis to include all participants with a bone age radiograph at screening. This analysis was performed after the clinical study report was completed & is included to match the FDA package insert.
Time Frame: Baseline to Month 6
Population: The baseline time frame was increased from the secondary outcome to this analysis to include all participants with a bone age radiograph at screening. This analysis was performed post hoc to match the FDA package insert.
Measure: Number; unit: Percentage of Participants
Groups:
- Leuprolide Acetate 11.25 mg: All subjects from both treatment groups who received 11.25 mg leuprolide acetate, both treatment naive and previously treated, were combined.
- Leuprolide Acetate 30 mg: All subjects from both treatment groups who received 30 mg leuprolide acetate, both treatment naive and previously treated, were combined.
Arm/Group | Leuprolide Acetate 11.25 mg | Leuprolide Acetate 30 mg
Number analyzed (Participants) | 33 | 40
Percentage of Participants | 87.9 | 75.0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were defined as any event with an onset data after the first dose of study drug and with an onset date no more than 30 days after the last day of study drug treatment which is 84 days after the last injection date.
Description: Safety analyses were performed with available data from all subjects who received at least 1 injection of study drug.
Arm/Group | Leuprolide Acetate 11.25 mg - Treatment Naive | Leuprolide Acetate 11.25 mg - Previous Treatment | Leuprolide Acetate 30 mg - Treatment Naive | Leuprolide Acetate 30 mg - Previous Treatment
Serious Adverse Events (participants affected / at risk) | 1/21 | 0/21 | 0/21 | 1/21
Other Adverse Events (participants affected / at risk) | 13/21 | 18/21 | 15/21 | 17/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Leuprolide Acetate 11.25 mg - Treatment Naive (N=21) | Leuprolide Acetate 11.25 mg - Previous Treatment (N=21) | Leuprolide Acetate 30 mg - Treatment Naive (N=21) | Leuprolide Acetate 30 mg - Previous Treatment (N=21)
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Weight Decreased (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Leuprolide Acetate 11.25 mg - Treatment Naive (N=21) | Leuprolide Acetate 11.25 mg - Previous Treatment (N=21) | Leuprolide Acetate 30 mg - Treatment Naive (N=21) | Leuprolide Acetate 30 mg - Previous Treatment (N=21)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1 | 0 | 2
Ear Pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 2
Goiter (Endocrine disorders) | 0 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 4 | 1
Injection Site Pain (General disorders) | 4 | 4 | 4 | 7
Pyrexia (General disorders) | 2 | 2 | 2 | 6
Ear Infection (Infections and infestations) | 0 | 2 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 2 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 4 | 1 | 1
Otitis Media (Infections and infestations) | 2 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 3 | 3 | 2
Arthropod Bite (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Weight Increased (Investigations) | 1 | 2 | 2 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 0
Headache (Nervous system disorders) | 1 | 4 | 6 | 6
Mood Altered (Psychiatric disorders) | 2 | 1 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 2 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2
Respiratory Disorders (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.